CLINICAL TRIAL: NCT02746887
Title: Risk Factors Related to Metabolic Syndrome in School-aged Children Who Were Born Preterm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung Han Shin, Professor, Seoul National University Hospital
Other Study IDs: 1509-030-702
Record Dates: First submitted 2015-12-09; First posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Preterm cohort: Preterm infants with a gestational age less than 32 weeks or birth weight less than 1,500 g
  Interventions: Other: Preterm/term cohort
- Term control cohort: Healthy term infants
  Interventions: Other: Preterm/term cohort

INTERVENTIONS:
Other: Preterm/term cohort

SUMMARY:
This is a follow-up cohort study of 8 years old children born preterm at Seoul National University Children's Hospital in Korea from 2008-2009.

The children will visit outpatient clinics for examinations regarding growth, obesity and other risk factors related to metabolic syndrome.

The purpose of this study is to compare growth and risk factors of metabolic syndrome among children born preterm and children born healthy term at school age

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infants and/or born less than 32 weeks of gestation age
* Healthy term infants for control group
* Parents and children accept of participation

Exclusion Criteria:

* Major congenital anomalies
* Neuromuscular disease
* Chromosomal anomalies
* Patients receiving growth hormone therapy
* Primary hypothyroidism

Ages: 8 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. school aged children who were born preterm with a gestational age less than 32 weeks or a birth weight less than 1,500 g
  2. school aged children who were born healthy term
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
number of participants with abnormal laboratory values and/or abnormal physical status | at 8 years corrected age

SECONDARY OUTCOMES:
The number of participants with catch-up growth failure | at 8 years corrected age
The number of participants with hypertension | at 8 years corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Seung Han Y Shin, MD, Principal Investigator — Seoul National University Children's Hospital
Locations (1):
- Seung Han Shin, Seoul, South Korea